CLINICAL TRIAL: NCT01584232
Title: A Phase 3 Study of LY2189265 Compared to Insulin Glargine in Patients With Type 2 Diabetes Mellitus on a Sulfonylurea and/or Biguanide
Brief Title: A Study of Dulaglutide in Japanese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14359; H9X-JE-GBDY (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-04-23; First posted 2012-04-24 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glucagon-like peptide-1 (GLP-1)
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Insulin Glargine; Sulfonylurea Compounds; Biguanides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2189265 + OAM (Experimental): LY2189265: 0.75 milligrams (mg), administered subcutaneously (SC), once weekly for 26 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of oral antihyperglycemic medication (OAM) throughout the study. OAMs included sulfonylureas (SU; glibenclamide, gliclazide, or glimepiride) and/or biguanides (BG; metformin or buformin).
  Interventions: Drug: LY2189265; Drug: Sulfonylureas (SU); Drug: Biguanide (BG)
- Insulin glargine + OAM (Active Comparator): Insulin glargine: dose based on targeting fasting blood glucose ≤110 milligrams per deciliter (mg/dL), administered subcutaneously (SC), once daily for 26 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of oral antihyperglycemic medication (OAM) throughout the study. OAMs included sulfonylureas (SU; glibenclamide, gliclazide, or glimepiride) and/or biguanides (BG; metformin or buformin).
  Interventions: Drug: Insulin glargine; Drug: Sulfonylureas (SU); Drug: Biguanide (BG)

INTERVENTIONS:
Drug: LY2189265
  Other Names: Dulaglutide
  Arms: LY2189265 + OAM
Drug: Insulin glargine
  Arms: Insulin glargine + OAM
Drug: Sulfonylureas (SU)
Drug: Biguanide (BG)

SUMMARY:
The purpose of this trial is to examine the efficacy and safety of once-weekly LY2189265 (dulaglutide) in participants with type 2 diabetes mellitus taking an oral antihyperglycemic medication (OAM).

DETAILED DESCRIPTION:
Rescue therapy (defined as alternative antihyperglycemic medication use or dose modification of oral antihyperglycemic medication [OAM]) may have been initiated during the planned treatment period if the participant discontinued study drug or met prespecified thresholds for severe, persistent hyperglycemia. Efficacy data, as well as data for hypoglycemic episodes from participants who permanently discontinued study treatment but switched to another diabetes medication and remained in the study, were censored from the point of initiating new treatment onwards.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have had a diagnosis of type 2 diabetes mellitus for at least 6 months before screening
* Participants who have been taking sulfonylurea (glibenclamide, gliclazide, or glimepiride) and/or biguanide (metformin or buformin). The dose of the drug(s) during the 8 weeks before screening must be stable
* Participants who have a qualifying glycosylated hemoglobin (HbA1c) value of 7.0% to 10.0% at screening
* Participants who have a body mass index (BMI) of 18.5 to 35.0 kilograms per meter squared (kg/m^2)

Exclusion Criteria:

* Participants who have a diagnosis of type 1 diabetes
* Participants who have previously been treated with any other glucagon-like peptide 1 (GLP-1) analog
* Participants who have received therapy with an alpha-glucosidase inhibitor (a-GI), thiazolidinedione (TZD), glinide, or dipeptidyl peptidase-IV (DPP-IV) inhibitor within 3 months before screening
* Participants who have been currently taking insulin or have had previous insulin treatment within 3 months before screening
* Participants who have obvious clinical signs or symptoms of pancreatitis, a history of chronic pancreatitis, or acute pancreatitis at screening, as determined by the investigator. Participants who have a serum amylase concentration ≥ 3 times the upper limit of the reference range and/or a serum lipase concentration ≥ 2 times the upper limit of the reference range, as determined by the central laboratory at screening
* Participants who have self or family history of medullary C-cell hyperplasia, focal hyperplasia, or medullary thyroid carcinoma (MTC)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- Japan (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kumamoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi

REFERENCES:
- [Derived] Suzuki S, Oura T, Takeuchi M, Boye KS. Evaluation of the impact of once weekly dulaglutide on patient-reported outcomes in Japanese patients with type 2 diabetes: comparisons with liraglutide, insulin glargine, and placebo in two randomized studies. Health Qual Life Outcomes. 2017 Jun 12;15(1):123. doi: 10.1186/s12955-017-0696-7. PMID 28606095

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LY2189265 + OAM | Insulin Glargine + OAM
Started | 181 | 180
Received at Least 1 Dose of Study Drug | 181 | 180
Completed | 173 | 177
Not Completed | 8 | 3
Not completed — Adverse Event | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of LY2189265 or insulin glargine.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2189265 + OAM | Insulin Glargine + OAM | Total
Number analyzed (Participants) | 181 | 180 | 361
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.52 (10.48) | 56.14 (11.33) | 56.83 (10.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 47 | 103
  Male | 125 | 133 | 258
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 181 | 180 | 361
Region of Enrollment [Number; unit: participants]
  Japan | 181 | 180 | 361

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at 26 Weeks
Description: Least squares (LS) means were calculated using a mixed-effects model for repeated measures (MMRM) analysis with treatment, visit, treatment-by-visit, oral antihyperglycemic medication regimen (sulfonylureas only, biguanides only, or both), and baseline body mass index (BMI) group (<25 or >=25 kilograms per meter squared [kg/m^2]) as fixed effects, baseline HbA1c as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or insulin glargine with evaluable HbA1c data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- LY2189265 + OAM: LY2189265: 0.75 mg, administered subcutaneously (SC), once weekly for 26 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of oral antihyperglycemic medication (OAM) throughout the study. OAMs included sulfonylureas (SU; glibenclamide, gliclazide, or glimepiride) and/or biguanides (BG; metformin or buformin).
Arm/Group | LY2189265 + OAM | Insulin Glargine + OAM
Number analyzed (Participants) | 178 | 179
percentage of HbA1c | -1.44 (0.05) | -0.90 (0.05)
Statistical Analysis 1: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Approximately 360 participants were to be randomized in a 1:1 ratio to LY2189265 or insulin glargine (IG). Assuming no difference in HbA1c change from baseline at Week 26 between LY2189265 and IG, this sample size would provide approximately 90% power to confirm non-inferiority of LY2189265 to IG. This computation was based on a non-inferiority margin of 0.4% with a standard deviation of 1.1%, a 1-sided alpha level of 0.025, and an 11% dropout rate between randomization and Week 26; Test type: Non-Inferiority or Equivalence — If the upper limit of the 95% Confidence Interval (CI) was <0.4%, then LY2189265 was declared non-inferior to insulin glargine. If the upper limit of the 95% CI was <0.0%, then LY2189265 was declared superior to insulin glargine; p < 0.001, Mixed Models Analysis — P-value is from the pairwise comparison of LS means using a mixed effects model with repeated measurements (MMRM); LS Mean Difference = -0.54, 95% CI 2-sided [-0.67 to -0.41]

2. Secondary Outcome: Percentage of Participants Who Achieved Glycosylated Hemoglobin (HbA1c) <=6.5% or <7% at 26 Weeks
Description: The percentage of participants achieving HbA1c level less than 7.0% and less than or equal to 6.5% was analyzed with a longitudinal logistic regression model with treatment, visit, treatment-by-visit, oral antihyperglycemic medication regimen (sulfonylureas only, biguanides only, or both), and baseline body mass index (BMI) group (<25 or >=25 kilograms per meter squared [kg/m^2]) as fixed effects, baseline HbA1c as a covariate, and participant as a random effect.
Time Frame: Up to 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or insulin glargine with evaluable HbA1c data. Only pre-rescue measurements were used. Missing endpoints were imputed with the last observation carried forward (LOCF), using only postbaseline data.
Measure: Number; unit: percentage of participants
Arm/Group | LY2189265 + OAM | Insulin Glargine + OAM
Number analyzed (Participants) | 178 | 179
percentage of participants
  HbA1c <=6.5% | 51.1 | 24.0
  HbA1c <7% | 71.3 | 45.8
Statistical Analysis 1: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c <=6.5%
Statistical Analysis 2: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Treatment comparison for HbA1c <7%

3. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG) at 26 Weeks
Description: Least squares (LS) means were calculated using a mixed-effects model for repeated measures (MMRM) analysis with treatment, visit, treatment-by-visit, oral antihyperglycemic medication regimen (sulfonylureas only, biguanides only, or both), and baseline body mass index (BMI) group (<25 or >=25 kilograms per meter squared [kg/m^2]) as fixed effects, baseline FBG as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or insulin glargine with evaluable fasting blood glucose data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2189265 + OAM | Insulin Glargine + OAM
Number analyzed (Participants) | 176 | 176
milligrams per deciliter (mg/dL) | -34.3 (1.9) | -37.8 (1.9)
Statistical Analysis 1: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p = 0.183, Mixed Models Analysis; LS Mean Difference = 3.5, 95% CI 2-sided [-1.7 to 8.7]

4. Secondary Outcome: Change From Baseline in 8-Point Self-Monitored Blood Glucose (SMBG) at 26 Weeks
Description: Participants were to test and record SMBG concentrations in their study diaries before each meal (breakfast, lunch, and dinner), approximately 2 hours after the start of each meal, at bedtime, and before breakfast the next morning (second pre-morning meal). Least squares (LS) means were calculated using analysis of covariance (ANCOVA) model with treatment, oral antihyperglycemic medication regimen (sulfonylureas only, biguanides only, or both), and baseline body mass index (BMI) group (<25 or >=25 kilograms per meter squared [kg/m^2]) as fixed effects and baseline SMBG as a covariate.
Time Frame: Baseline, Up to 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or insulin glargine with evaluable SMBG data. Only pre-rescue measurements were used. Missing endpoints were imputed with the last observation carried forward (LOCF), using only postbaseline data.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | LY2189265 + OAM | Insulin Glargine + OAM
Number analyzed (Participants) | 178 | 179
milligrams per deciliter (mg/dL)
  Pre-morning meal (n=178, 179) | -33.49 (1.65) | -38.66 (1.64)
  2 hours post-morning meal (n=178, 179) | -49.54 (3.33) | -36.14 (3.31)
  Pre-midday meal (n=178, 179) | -36.16 (2.68) | -27.94 (2.66)
  2 hours post-midday meal (n=178, 179) | -43.51 (3.27) | -20.30 (3.25)
  Pre-evening meal (n=178, 179) | -31.14 (2.77) | -17.50 (2.75)
  2 hours post-evening meal (n=177, 178) | -46.68 (3.05) | -15.55 (3.03)
  Bedtime (n=177, 172) | -41.53 (2.95) | -17.79 (2.96)
  Second pre-morning meal (n=178, 179) | -30.81 (1.60) | -37.02 (1.59)
Statistical Analysis 1: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p = 0.022, ANCOVA — Treatment comparison for pre-morning meal; LS Mean Difference = 5.16, 95% CI 2-sided [0.76 to 9.56]
Statistical Analysis 2: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p = 0.003, ANCOVA — Treatment comparison for 2 hours post-morning meal; LS Mean Difference = -13.40, 95% CI 2-sided [-22.28 to -4.52]
Statistical Analysis 3: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p = 0.025, ANCOVA — Treatment comparison for pre-midday meal; LS Mean Difference = -8.22, 95% CI 2-sided [-15.37 to -1.06]
Statistical Analysis 4: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison for 2 hours post-midday meal; LS Mean Difference = -23.22, 95% CI 2-sided [-31.92 to -14.51]
Statistical Analysis 5: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison for pre-evening meal; LS Mean Difference = -13.63, 95% CI 2-sided [-21.03 to -6.24]
Statistical Analysis 6: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison for 2 hours post-evening meal; LS Mean Difference = -31.13, 95% CI 2-sided [-39.26 to -23.00]
Statistical Analysis 7: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p < 0.001, ANCOVA — Treatment comparison for bedtime; LS Mean Difference = -23.73, 95% CI 2-sided [-31.68 to -15.79]
Statistical Analysis 8: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p = 0.005, ANCOVA — Treatment comparison for second pre-morning meal; LS Mean Difference = 6.21, 95% CI 2-sided [1.92 to 10.50]

5. Secondary Outcome: Change From Baseline in Body Weight at 26 Weeks
Description: Least squares (LS) means were calculated using a mixed-effects model for repeated measures (MMRM) analysis with treatment, visit, treatment-by-visit, oral antihyperglycemic medication regimen (sulfonylureas only, biguanides only, or both), and baseline body mass index (BMI) group (<25 or >=25 kilograms per meter squared [kg/m^2]) as fixed effects, baseline body weight as a covariate, and participant as a random effect.
Time Frame: Baseline, 26 weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or insulin glargine with evaluable body weight data. Only pre-rescue measurements were used.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2189265 + OAM | Insulin Glargine + OAM
Number analyzed (Participants) | 180 | 180
kilograms (kg) | -0.48 (0.17) | 0.94 (0.17)
Statistical Analysis 1: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.42, 95% CI 2-sided [-1.89 to -0.94]

6. Secondary Outcome: Percentage of Participants With Hypoglycemic Episodes
Description: The percentage of participants with hypoglycemic episodes was calculated by dividing the number of participants with at least one hypoglycemic episode over the 26-week treatment period by the total number of participants analyzed, multiplied by 100%. All classifications of hypoglycemia (documented symptomatic, asymptomatic, severe, nocturnal, non-nocturnal, probable symptomatic, relative, and unspecified) were included, except for episodes of relative hypoglycemia that were not severe. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 Weeks
Population: Participants who were randomized and received at least 1 dose of LY2189265 or insulin glargine. Only pre-rescue data was used.
Measure: Number; unit: percentage of participants
Arm/Group | LY2189265 + OAM | Insulin Glargine + OAM
Number analyzed (Participants) | 181 | 180
percentage of participants | 26.0 | 47.8
Statistical Analysis 1: Comparison: LY2189265 + OAM vs Insulin Glargine + OAM; Test type: Superiority or Other; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Arm/Group | LY2189265 + OAM | Insulin Glargine + OAM
Serious Adverse Events (participants affected / at risk) | 9/181 | 3/180
Other Adverse Events (participants affected / at risk) | 133/181 | 111/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2189265 + OAM (N=181) | Insulin Glargine + OAM (N=180)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Spinal cord infarction (Nervous system disorders) | 0 (0) | 1 (1)
Viith nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2189265 + OAM (N=181) | Insulin Glargine + OAM (N=180)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 1 (1)
Cystoid macular oedema (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 4 (4) | 2 (2)
Dry eye (Eye disorders) | 1 (1) | 1 (1)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 1 (2)
Retinal vein occlusion (Eye disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (13) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (6) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 16 (19) | 6 (7)
Dental caries (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 22 (31) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (6) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastritis atrophic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (27) | 2 (2)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 9 (13) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Infusion site induration (General disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (1)
Injection site dermatitis (General disorders) | 1 (21) | 0 (0)
Injection site hypersensitivity (General disorders) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (2)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema due to renal disease (General disorders) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic calcification (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3) | 3 (3)
Seasonal allergy (Immune system disorders) | 1 (1) | 2 (2)
Abscess oral (Infections and infestations) | 1 (1) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 7 (10)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 0 (0)
Enteritis infectious (Infections and infestations) | 2 (2) | 2 (2)
Enterocolitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 3 (3)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 6 (6) | 2 (2)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lymphadenitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 49 (55) | 46 (57)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (4) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 2 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 4 (6)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 3 (3) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 9 (9) | 1 (1)
Occult blood (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (8) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Vith nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Alcohol problem (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 2 (2) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 2 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/125 (1) | 1/133 (1)
Endometriosis (Reproductive system and breast disorders) | 1/56 (1) | 0/47 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Asteatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (5)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days